CLINICAL TRIAL: NCT05161325
Title: An Observational Study of Effectiveness and Safety of the First-Line Nivolumab Plus Ipilimumab With or Without Chemotherapy for Advanced/Recurrent Non-Small Cell Lung Cancer in Japan
Brief Title: A Study of Effectiveness and Safety of the First-Line Nivolumab Plus Ipilimumab With or Without Chemotherapy for Advanced/Recurrent Non-Small Cell Lung Cancer in Japan
Acronym: LIGHT-NING
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharma USA Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-64A
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: BMS-936558; ONO-4538; Nivolumab; Ipilimumab; Retrospective; Observational
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort 1: Participants with untreated advanced or recurrent non-small cell lung cancer (NSCLC) receiving first-line nivolumab plus ipilimumab with or without chemotherapy

SUMMARY:
The purpose of this observational study is to assess the effectiveness and safety of Nivolumab plus Ipilimumab with or without chemotherapy as first-line treatment for participants with untreated advanced or recurrent NSCLC in the real world setting in Japan.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed advanced or recurrent NSCLC
* Participants who have received or scheduled to administrate nivolumab plus ipilimumab with or without chemotherapy as first-line treatment from the date of approval of nivolumab plus ipilimumab with or without chemotherapy to November 30, 2021.

  1. Pemetrexed plus cisplatin or carboplatin for participants with non- squamous histology and paclitaxel plus carboplatin for participants with squamous histology are only acceptable combinations of chemotherapy.

Exclusion Criteria:

* In participants with non-squamous histology, participants who are confirmed to be positive for EGFR gene mutation or ALK fusion gene for which EGFR tyrosine kinase inhibitor or ALK tyrosine kinase inhibitor is indicated.
* Participants who had antineoplastic treatment as first-line treatment of advanced or recurrent NSCLC prior to initiation of nivolumab plus ipilimumab with or without chemotherapy.

However, participants who correspond to a) or b) below will be included in this study.

1. Prior perioperative chemotherapy or Stage III chemoradiotherapy or durvalumab combination chemoradiotherapy.
2. Participants who are received or have received bisphosphonates or denosumab for bone metastasis

   * Participants who initiated treatment with nivolumab plus ipilimumab and added chemotherapy from the second course onwards.
   * Participants who received investigational anti-tumor drug in clinical trial after being diagnosed with NSCLC
   * Other participants who are judged by the investigators to be inappropriate for enrollment in this study

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a descriptive study of participants who received nivolumab plus ipilimumab with or without chemotherapy within 1 year of approval. In this study, the target sample size is set at 500 participants based on the feasibility to investigate the actual clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Duration of treatment | Up to 1 year
  Time from the initiation date of nivolumab plus ipilimumab with or without chemotherapy among eligible participants to the last date of treatment as an event.
Rates of participants with second-line treatment | Up to 1 year
  The rate of eligible participants who have completed nivolumab plus ipilimumab with or without chemotherapy during the observation period and have initiated second-line treatment
Overall survival (OS) | Up to 1 year
  Defined as the time between the date of initiation of nivolumab plus ipilimumab with or without chemotherapy and the date of death from any cause among eligible participants.
Incidence of Common Terminology Criteria for Adverse Events (CTCAE) v 5.0 Grade 3 or higher immune-related adverse events [irAEs] | Up to 1 year
Time to next treatment [(TNT) | Up to 1 year
  Defined as the time between the date of combination therapy with nivolumab plus ipilimumab with or without chemotherapy initiation among eligible participants and the date of second-line treatment initiation or the date of death from any cause, whichever occurs first.
Treatment-free survival (TFS) | Up to 1 year
  Defined as the time between the date of nivolumab plus ipilimumab with or without chemotherapy cessation among eligible participants and the date of second-line treatment initiation or the date of death from any cause, whichever occurs first.
Treatment continuation rate | Up to 1 year
  The rate of eligible participants who have continued nivolumab plus ipilimumab with or without chemotherapy during the observation period.
Incidence of treatment-related adverse events (TRAEs) leading to treatment discontinuation | Up to 1 year

SECONDARY OUTCOMES:
Progression-free survival (PFS) in participants assessed for tumor response according to RECIST v 1.1 | Up to 1 year
Objective response rate (ORR) in participants evaluated for tumor response according to RECIST v 1.1 | Up to 1 year
Disease control rate (DCR) in participants evaluated for response in accordance with RECIST v 1.1 | Up to 1 year
Duration of response (DOR) in participants evaluated for tumor response in accordance with RECIST v 1.1 | Up to 1 year
Overall Survival (OS) by patient background | Up to 1 year
Time to next treatment (TNT) by patient background | Up to 1 year
Treatment-free survival (TFS) by patient background | Up to 1 year
Treatment continuation rate by patient background | Up to 1 year
Incidence of CTCAE v 5.0 Grade 3 or higher irAEs by patient background | Up to 1 year
Incidence of TRAEs leading to treatment discontinuation by patient background | Up to 1 year
Overall survival of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Time to next treatment of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Treatment-free survival of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Treatment continuation rate of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Incidence of CTCAE v 5.0 Grade 3 or higher irAEs of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Incidence of TRAEs leading to treatment discontinuation of nivolumab plus ipilimumab with or without chemotherapy by adjustment for confounding factors | Up to 1 year
Time to onset of immune-related adverse events (irAEs) to be collected, treatment for these events and time to symptom improvement, and impact on effectiveness | Up to 1 year
Duration of treatment of second-line treatment | Up to 1 year
Reasons for treatment discontinuation of second-line treatment | Up to 1 year
Treatment related death of second-line treatment | Up to 1 year
Response rate of second-line treatment | Up to 1 year
Overall survival in participants who discontinued treatment due to treatment-related adverse events within 90 days | Up to 1 year
Time to next treatment in participants who discontinued treatment due to treatment-related adverse events within 90 days | Up to 1 year
Treatment-free survival in participants who discontinued treatment due to treatment-related adverse events within 90 days | Up to 1 year
Treatment continuation rate in participants who discontinued treatment due to treatment-related adverse events within 90 days | Up to 1 year
Duration of treatment of second-line treatment in participants with disease progression within 90 days | Up to 1 year
Reasons for treatment discontinuation of second-line treatment in participants with disease progression within 90 days | Up to 1 year
Overall survival of second-line treatment in participants with disease progression within 90 days | Up to 1 year
Response rate of second-line treatment in participants with disease progression within 90 days | Up to 1 year
Treatment related death of second-line treatment in participants with disease progression within 90 days | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Minato-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm